CLINICAL TRIAL: NCT02991651
Title: A Phase I Study of IRX4204 in Combination With Erlotinib in Patients With Previously Treated Advanced Non-Small Cell Lung Cancer
Brief Title: Study of IRX4204 With Erlotinib in Previously Treated Advanced NSCLC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study drug supply expired. No replacement manufactured. Sponsor did not want to continue study.
Sponsor: Io Therapeutics (Industry)
Collaborators: Dartmouth College (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRX4204 NSCLC 1 01 2015
Record Dates: First submitted 2016-12-07; First posted 2016-12-13 (Estimated); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer, Nonsmall Cell
Keywords: RXR agonist IRX4204 erlotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — IRX4204; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose Level 1 (Experimental): IRX4204 5 mg/day PO + erlotinib 100 mg/day PO
  Interventions: Drug: IRX4204; Drug: erlotinib
- Dose Level 2 (Experimental): IRX4204 5 mg/day PO + erlotinib 150 mg/day PO
  Interventions: Drug: IRX4204; Drug: erlotinib
- Dose Level 3 (Experimental): IRX4204 10 mg/day PO + erlotinib 150 mg/day PO
  Interventions: Drug: IRX4204; Drug: erlotinib

INTERVENTIONS:
Drug: IRX4204 — RXR agonist
Drug: erlotinib — inhibitor of phosphorylation of the tyrosine kinase associated with the epidermal growth factor receptor

SUMMARY:
Patient selection: a) Pathological confirmation of non-small cell lung cancer without activating EGFR mutations; b) Advanced stage disease (IV or IIIB with malignant effusion) with at least two prior chemotherapy regimens; c) No available curative therapy; d) Pregnant women are excluded; e) Informed consent.

Pretreatment evaluation: a) Medical history and physical examination; b) Hepatic and renal function (bilirubin, aspartate aminotransaminase, creatinine); c) Preoperative staging evaluation including CT-chest or PET/CT scan;

Treatment plan: Three dose levels of IRX4204 and erlotinib will be studied using intra-patient dose escalation for dose levels 1 and 2. These study agents will be administered orally until progression of disease, unacceptable toxicities, activation of a phase II study of the combination, or exhaustion of the IRX4204 drug supply.

Evaluation on study: Adverse events will be graded on a scale of 0 to 5, using the Common Terminology Criteria for Adverse Events (CTCAE) v. 4.0. Efficacy will be assessed using the RECIST v1.1 criteria based on CT-chest or PET/CT scan after 8 weeks of study treatment.

DETAILED DESCRIPTION:
Numerous studies in pre-clinical models and in human clinical trials have clearly established the potential for the use of rexinoids in the treatment and prevention of cancer. IRX4204, a second generation rexinoid, is a highly potent and specific activator of RXRs. Because IRX4204 is significantly more potent and more selective for the RXRs relative to the RARs than a first generation approved RXR agonist drug, bexarotene, it potentially will be associated with fewer adverse events and greater activity in clinical use. Preclinical studies of the combination of IRX4204 plus erlotinib, and previous clinical studies of the combination of the bexarotene plus erlotinib indicated at least additive beneficial effects for treatment of NSCLC. This study seeks to investigate the safety and activity of IRX4204 in combination with erlotinib in patients with previously treated advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed stage IV non-small cell lung cancer, or recurrent non-small cell lung cancer which is not amenable to curative intent therapy.
* Documented disease progression on at least two prior lines of chemotherapy for advanced NSCLC. Progression within 6 months of adjuvant chemotherapy or definitive chemoradiation will count as one line of therapy.
* Age ≥18 years.
* ECOG performance status ≤2.
* Ability to take pills by mouth.
* Patients must have normal organ and marrow function as defined below:
* Leukocytes ≥3,000/mcL
* Absolute neutrophil count ≥1,500/mcL
* Platelets ≥100,000/mcL
* Hemoglobin ≥8.5 g/dL
* Total bilirubin ≤1.5 x institutional upper limit of normal (ULN)
* AST(SGOT)/ALT(SGPT) ≤2.5 × ULN or ≤5 x ULN if metastases to the liver
* Creatinine clearance ≥40 mL/min
* Patients with asymptomatic brain metastases are allowed, as long as they are stable and do not require treatment with anticonvulsants or escalating doses of steroids. Maximum daily dose of steroids should be prednisone 20 mg or equivalent. Radiation therapy for brain metastases must be completed at least 14 days prior to treatment on protocol.
* Women of child-bearing potential and men must agree to use highly effective contraception (if using hormonal birth control must add a second barrier method; abstinence) prior to study entry, for the duration of study participation as well as for at least 1 month after the last dose of IRX4204. Men treated or enrolled on this protocol must also agree to use highly effective contraception prior to the study, for the duration of study participation and 3 months after completion of IRX4204 administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study.
* Activating EGFR mutations detected in the tumor.
* Prior treatment with an EGFR tyrosine kinase inhibitor.
* Prior treatment with IRX4204 or another retinoid or rexinoid administered for the purpose of cancer treatment. Prior topical retinoid use is allowed.
* History of allergic reactions attributed to IRX4204 or erlotinib or to compounds of similar chemical or biologic composition.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and nursing women.
* Patients with a history of another active malignancy within the past two years, with the exception of non-melanoma cutaneous malignancy, cervical carcinoma in situ, or ductal carcinoma in situ which has been successfully treated with curative intent therapy.
* Any gastrointestinal disorder expected to limit absorption of IRX4204 or erlotinib.
* Patients with a history of active thyroid disease. However, patients with a history of hypothyroidism maintained in euthyroid state by supplementation with thyroid hormone, or a thyroid hormone containing preparation may be enrolled.
* Patients taking coumarin-derived anticoagulants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-12-07 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Safety of co-administration of IRX4204 + erlotinib to determine recommended phase 2 dose based on number of participants experiencing treatment-related adverse events as assessed as grade 4 by CTCAE v4.0 | 30 days
  To determine the recommended phase II dose (RP2D) for the combination of IRX4204 and erlotinib.

SECONDARY OUTCOMES:
toxicity profile of the combination of IRX4204 and erlotinib based on number of participants experiencing treatment-related grades 1-4 adverse events as assessed by CTCAE v4.0 | one month
disease control rate (defined as rate of stable disease + partial response + complete response) | six months
progression free survival (PFS) | six months
overall survival (OS) | six months
response rate by RECIST 1.1 | six months

CONTACTS AND LOCATIONS:
Overall Officials: Martin E Sanders, MD, Study Director — Io Therapeutics, Inc.
Locations (1):
- Geisel School of Medicine at Dartmouth, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No